CLINICAL TRIAL: NCT02215499
Title: A Double-Blind, Phase 1, Single-Center, Single-Ascending Dose Study of JZP-386 Compared to Xyrem® vs. Placebo to Evaluate the Safety and Pharmacokinetics
Brief Title: A Phase 1, Single Dose Study of JZP-386 to Evaluate Safety, Pharmacokinetics and Pharmacodynamics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CP386.1001
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Narcolepsy, Excessive Daytime Sleepiness
Keywords: JZP-386, Xyrem, sodium oxybate
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Xyrem® (Active Comparator): Oral suspension
  Interventions: Drug: Placebo; Drug: Sodium Oxybate
- JZP-386 (Experimental): Oral suspension
  Interventions: Drug: Placebo; Drug: JZP-386
- Placebo (Placebo Comparator): Oral suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
Drug: Sodium Oxybate
  Other Names: Xyrem®
  Arms: Xyrem®
Drug: JZP-386
  Arms: JZP-386

SUMMARY:
This study is being conducted to evaluate the safety, tolerability, blood distribution and effectiveness single ascending doses of JZP-386 compared to doses of Xyrem® and placebo.

DETAILED DESCRIPTION:
This is a Phase 1, single center, single-ascending dose, sequential, randomized, and crossover study.

Following a Screening period of up to 21 days, eligible subjects will be randomized different dosing sequences, with approximately 4 subjects allocated to each dosing sequence. The total in-clinic duration for each subject will be 24 days (including the admission day prior to the first dosing period).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteer subjects, 18 to 50 years of age, inclusive.

Exclusion Criteria:

Clinically significant history of unstable medical abnormality. Inability to cooperate with study procedures. Female subjects with a positive pregnancy test result, nursing or lactating. Participation in any other investigational drug trial within 90 days prior to screening. A history of prescription drug abuse, or illicit drug or known drug dependence within last 5 years prior to screening. Use of any prescription medication within 14 days prior to dosing. A history of alcohol abuse or dependence.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
safety | 3 days
  Evaluate and compare the safety including adverse event monitoring (number and type of events), vital signs, pulse oximetry of single ascending doses of JZP-386 to Xyrem (sodium oxybate) and placebo in healthy subjects.

SECONDARY OUTCOMES:
pharmacokinetics | 12 hours
  Evaluate the pharmacokinetics (AUC, Cmax) of of JZP-386 compared to Xyrem in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: LuAnn Sabounjian, Study Director — Concert Pharmaceuticals
Locations (1):
- Quotient Clinical Ltd., Ruddington, Nottingham, United Kingdom